CLINICAL TRIAL: NCT01301638
Title: Retrospective Evaluation of Safety and Efficacy of Daptomycin Used in Patients With Serious Gram-positive Infections
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Department of Internal Medicine, Section of Infectious Disease, Far Eastern Memorial Hospital
Other Study IDs: 099150-E
Record Dates: First submitted 2011-02-21; First posted 2011-02-23 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2011-02

CONDITIONS: Bacteremia; Endocarditis; Serious Gram-positive Infections
MeSH Terms: conditions — Bacteremia; Endocarditis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Before Daptomycin (Cubicin ®) approved by the U.S. FDA in 2003, There were large-scale clinical trials conducted that included more than 1,000 subjects and than Daptomycin got complicated skin and soft tissue infections (CSSSI) indication. After 2004, Daptomycin got new indications about bacteremia and endocarditis due to success outcomes in the clinical trial which included infected in blood flow and endocardial infected patients.

All subjects in Daptomycin clinical trials are European and American race. It is necessary that collecting safety and efficacy data of Daptomycin in Taiwan race. I will intent to evaluate the safety and efficacy of Daptomycin which were used in patients with serious gram-positive infections retrospectively. And the outcome could be a reference for Daptomycin future using.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients who were prescribed daptomycin from 1st January 2009 to 31st December 2010 for gram positive infections as deemed necessary by his/her treating physician. And patients received Daptomycin therapy for at least 3 days.

Exclusion Criteria:

* Patients received Daptomycin therapy for over 3 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Before Daptomycin (Cubicin ®) approved by the U.S. FDA in 2003, There were large-scale clinical trials conducted that include more than 1,000 subjects and than Daptomycin got complicated skin and soft tissue infections (CSSSI) indication. After 2004, Daptomycin got new indications about bacteremia and endocarditis due to success outcomes in the clinical trial which included infected in blood flow and endocardial infected patients.
  All subjects in Daptomycin clinical trials are European and American race. It is necessary that collecting safety and efficacy data of Daptomycin in Taiwan race. I will intent to evaluate the safety and efficacy of Daptomycin which were used in patients with serious gram-positive infections retrospectively. And the outcome could be a reference for Daptomycin future using
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-02

CONTACTS AND LOCATIONS:
Overall Officials: Men_Shan Hsu, medicine, Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, Taipei, Taiwan, Taiwan